CLINICAL TRIAL: NCT02700672
Title: Predicting Falls Among Institutionalized and Non-institutionalized Older Adults: The Role of Cognition and Gait Speed
Brief Title: Influence of Cognition and Gait on Falls
Acronym: ICGF
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Jose Carlos Fernandes Galduroz MD, Principal Investigator, Federal University of São Paulo
Other Study IDs: Falls&Cognition&Gait
Record Dates: First submitted 2016-01-07; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Accidental Falls
Keywords: Ageing; Cognition; Executive Function; Gait
MeSH Terms: interventions — Observation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Institutionalized older adults: Observational study
  Interventions: Other: Observational study
- Non-institutionalized older adults: Observational study
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study: kinematic variables, falls and executive function were analyzed

SUMMARY:
The study analyses if cognition and gait speed can predict falls in a community-dwelling people and ambulant long term care residents

DETAILED DESCRIPTION:
Falls are some of the most common events among elderly people. The odds of recurrent falls increase every year, which can cause impairment in basic activities of daily living, social isolation, fear of falling again and death. The aim of the present study is to analyze the role of cognition and gait speed as predictors to falls in institutionalized and non-institutionalized elderly people.

Methods:Twenty-five individuals living in a long-term care facility and 25 non-institutionalized individuals participated in the study. A questionnaire about their history of falls, tests to evaluate cognition (global and executive function) and a pedometer with an accelerometer to measure kinematic variables were applied.

ELIGIBILITY:
Inclusion Criteria:

* People who could walk with or without ambulation devices
* Mini-Mental State Examination score according to schooling

Exclusion Criteria:

* Terminal illnesses
* Bedridden
* Unable to see or hear
* Use of benzodiazepines

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty-five individuals living in a long term care facility and twenty-five older adults from community
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cognitive predictor of falls assessed with the Mini-Mental State Examination | falls on past 12 months
  To measure cognitive predictor will be used Mini-Mental State Examination

SECONDARY OUTCOMES:
Executive function predictor of falls assessed with the Wisconsin Card Sort Test | falls on past 12 months
  To measure executive function will be used Wisconsin Card Sort Test
Gait speed predictor of falls assessed with an accelerometer | falls on past 12 months
  To measure gait speed will be used an accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Galduróz, PhD, Principal Investigator — Federal University of São Paulo